CLINICAL TRIAL: NCT00175682
Title: Prophylactic Value of Prazosin in Reducing the Objective and Subjective Measures of Autonomic Dysreflexia Provoked by Ejaculation in Men With Spinal Cord Injury
Brief Title: Prazosin Vibrostimulation Autonomic Dysreflexia and Spinal Cord Injury Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: C04-0343
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Autonomic Dysreflexia
Keywords: Autonomic Dysreflexia; SCI; Vibrostimulation; Ejaculation
MeSH Terms: conditions — Autonomic Dysreflexia | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Prazosin HCL — See Detailed Description

SUMMARY:
Sexuality is a high rehabilitative priority for persons following a spinal cord injury (SCI). Sexual acts can lead to autonomic dysreflexia (AD), dangerous consequences such as a sudden increase in blood pressure, severe headache, sweating above the level of the lesion and low heart rate to name a few. Ejaculation in men can provoke these significant symptoms and therefore men and women may refrain from a sexual life and biological parenthood. Adalat is the most common antihypertensive used in fertility clinics to reduce the incidence of AD. It dramatically reduces blood pressure and, therefore, results in side effects such as dizziness, fatigue and weakness. The investigators hypothesize that Minipress® (prazosin HCL), a blood pressure medication, which has a slower and less abrupt suppressive effect on blood pressure, would be a safe, effective and more appropriate medication for use in the outpatient sperm retrieval clinic and potentially for private use.

DETAILED DESCRIPTION:
The consequences of sexual activity in the spinal cord injured (SCI) population include responses beyond the voluntary control of the person with SCI such as bladder and bowel issues, spasms and autonomic dysreflexia (AD). Currently we are looking at predictive measurements for AD during ejaculation in a controlled setting. Immediate-release Nifedipine (Adalat), a well-known medication used for the treatment of AD is the most commonly prescribed prophylactic antihypertensive used in sperm retrieval and urological procedures. Nifedipine has rapid onset (minutes) and dramatically lowers blood pressure for periods of up to five hours and results in dizziness, fatigue and weakness. As a sperm retrieval center not equipped for hypotensive resuscitation measures, we have refrained from using Nifedipine prior to procedures in hypotensive SCI men at risk for AD.

Our objective is to study the prophylactic capacity of a lesser prescribed antihypertensive medication Prazosin on its ability to reduce the objective and subjective measures of autonomic dysreflexia in order to assess its immediate potential for home use. Prazosin is an alpha-adrenergic blocker and has a slower and less abrupt suppressive effect on blood pressure. We hypothesize that it will reduce AD signs and symptoms, reduce the severity of cardiovascular changes, and improve client comfort without reduction in safety. Having 8 male subjects as their own controls, we plan to examine the objective (beat to beat blood pressure, EKG and visible body signs) and subjective (patient's symptomatic report) parameters of AD provoked by vibrostimulation and ejaculation on and off Minipress (Prazosin HCL). Statistical analysis will be done on three independent observations:

1. absolute blood pressure values and reduction in abnormal heart rhythms
2. signs and symptoms of AD
3. client confidence to undergo ejaculation

We will correlate objective parameters with the subjective findings to see if these observations can be predictive in determining the predictability and severity of AD and the effectiveness of Prazosin as prophylactic AD medication in an outpatient clinic or a private home setting during sexual activities.

ELIGIBILITY:
Inclusion Criteria:

* Male with spinal cord injured above level T6 of greater than one year's duration

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2004-12; Primary Completion 2011-07-28 (Actual); Study Completion 2011-07-28 (Actual)

PRIMARY OUTCOMES:
The hypothesis will be tested by measuring three parameters during prazosin and non-prazosin trials in which ejaculation occurs.
Objective parameters: absolute beat-to-beat BP, differences between systolic and diastolic BP readings, heart rate variability, heart rate and ECG readings (looking for irregular rhythms) and visible signs of AD experienced by the subject
Subjective parameters: subject perceived efficacy and side effects of the medication and willingness to use the medication at home

SECONDARY OUTCOMES:
Secondary outcomes will include the subject's knowledge of AD.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Elliott, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, BC Centre for Sexual Medicine, Vancouver, British Columbia, Canada